CLINICAL TRIAL: NCT04639219
Title: A Phase II, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of Trastuzumab Deruxtecan (T-DXd) for the Treatment of Unresectable and/or Metastatic Solid Tumors Harboring HER2 Activating Mutations Regardless of Tumor Histology
Brief Title: A Study of T-DXd for the Treatment of Solid Tumors Harboring HER2 Activating Mutations
Acronym: DPT01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D967MC00001; 2024-516158-22-00 (Other: EU-CTR Number); 2020-002368-30 (EudraCT Number)
Record Dates: First submitted 2020-10-26; First posted 2020-11-20 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors With HER2 Mutation,eg:Colorectal,Urothelial,Gastric, Hepatobiliary,Endometrial,Melanoma,Ovarian,Cervical,Salivary Gland,Pancreatic,Breast
Keywords: HER2; T-DXd; DS-8201a; Trastuzumab Deruxtecan; Metastatic; Solid Tumors; Histology Agnostic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Masking Description: None (open-label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-DXd (Experimental): T-DXd monotherapy
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan (T-DXd) by intravenous infusion
  Other Names: DS-8201a (T-DXd)

SUMMARY:
This is an open-label, multi-center, single arm, Phase II study to evaluate the efficacy and safety of T-DXd for the treatment of unresectable and/or metastatic solid tumors harboring specific HER2 activating mutations regardless of tumor histology. The target population are patients who have progressed following prior treatment or who have no satisfactory alternative treatment options, including approved second line therapies in the specific tumor type. Pre-specified HER2 mutations will be locally assessed using NGS tests or alternative methods. Prior HER2 targeting therapy is permitted.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old. Other age restrictions may apply as per local regulations.
* Unresectable and/or metastatic solid tumors with pre-specified HER2 mutations (S310F, S310Y, G660D, R678Q, D769Y, D769H, V777L, Y772_A775dup / A775_G776insYVMA, L755S, G778_P780dup / P780_Y781insGSP, T862A, and V842I locally determined by NGS or a validated nucleic acid-based methodology (eg, qPCR, digital PCR) on tumor tissue, who have progressed following prior treatment or who have no satisfactory alternative treatment options.
* Prior HER2 targeted therapy is permitted.
* All patients must provide an FFPE tumor sample for retrospective central HER2 testing.
* LVEF ≥50%
* ECOG 0-1
* All patients have measurable target disease assessed by the Investigator based on RECIST v1.1

Exclusion Criteria:

* HER2 overexpressing (IHC3+ or IHC2+/ISH+) breast, gastric or gastroesophageal junction adenocarcinoma.
* HER2 mutant NSCLC.
* Medical history of myocardial infarction within 6 months before randomization/enrolment, symptomatic CHF, unstable angina pectoris, clinically important cardiac arrhythmias, or a recent (< 6 months) cardiovascular event including stroke.
* History of non-infectious pneumonitis/ILD, current ILD, or where suspected ILD cannot be ruled out by imaging at screening
* Corrected QT interval by Fridericia's formula (QTcF) prolongation to > 470 msec (females) or > 450 msec (males) based on average of the screening triplicate 12-lead ECG.
* Lung-specific intercurrent clinically significant severe illnesses.
* History of active primary immunodeficiency, known HIV, active HBV or HCV infection
* Uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals
* Pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART).
* Has spinal cord compression or clinically active central nervous system metastases.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2026-07-14 (Estimated)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (9):
  - Research Site, Santa Rosa, California
  - Research Site, Muncie, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Middletown, New Jersey
  - Research Site, Commack, New York
  - Research Site, Harrison, New York
  - Research Site, New York, New York
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
- Research Site, Anderlecht, Belgium
- Research Site, Toronto, CA, Canada
- Research Site, Copenhagen, Denmark
- France (3):
  - Research Site, Bordeaux
  - Research Site, Lyon
  - Research Site, Villejuif
- Italy (2):
  - Research Site, Milan
  - Research Site, Napoli
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Suita-shi
- Research Site, Seoul, South Korea
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool .
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
  For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Li BT, Meric-Bernstam F, Bardia A, Naito Y, Siena S, Aftimos P, Anderson I, Curigliano G, de Miguel M, Kalra M, Oh DY, Park JO, Postel-Vinay S, Rha SY, Satoh T, Spanggaard I, Michelini F, Smith A, Machado KK, Saura C; DESTINY-PanTumor01 study group. Trastuzumab deruxtecan in patients with solid tumours harbouring specific activating HER2 mutations (DESTINY-PanTumor01): an international, phase 2 study. Lancet Oncol. 2024 Jun;25(6):707-719. doi: 10.1016/S1470-2045(24)00140-2. Epub 2024 May 3. PMID 38710187
- [Derived] Jhaveri K, Eli LD, Wildiers H, Hurvitz SA, Guerrero-Zotano A, Unni N, Brufsky A, Park H, Waisman J, Yang ES, Spanggaard I, Reid S, Burkard ME, Vinayak S, Prat A, Arnedos M, Bidard FC, Loi S, Crown J, Bhave M, Piha-Paul SA, Suga JM, Chia S, Saura C, Garcia-Saenz JA, Gambardella V, de Miguel MJ, Gal-Yam EN, Rapael A, Stemmer SM, Ma C, Hanker AB, Ye D, Goldman JW, Bose R, Peterson L, Bell JSK, Frazier A, DiPrimeo D, Wong A, Arteaga CL, Solit DB. Neratinib + fulvestrant + trastuzumab for HR-positive, HER2-negative, HER2-mutant metastatic breast cancer: outcomes and biomarker analysis from the SUMMIT trial. Ann Oncol. 2023 Oct;34(10):885-898. doi: 10.1016/j.annonc.2023.08.003. Epub 2023 Aug 18. PMID 37597578
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D967MC00001&attachmentIdentifier=fbe84ef4-bbba-4563-b487-fb52a7149bd6&fileName=d967mc00001-study-CSR_synopsis_Marked_for_redaction_Draft_2_Redacted_PDFA.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D967MC00001&attachmentIdentifier=adaa1038-46d9-4d78-b5f7-b20fb195c3e4&fileName=d967mc00001-sap-ed-3_DP-01_REDACTED_28Sep2023_PDFA.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D967MC00001&attachmentIdentifier=88099069-8e9a-490f-95a8-03c1a97112cb&fileName=d967mc00001-csp-v1_DP-01_REDACTED_28Sep2023_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II multicenter, open-label study was conducted in participants with unresectable and/or metastatic solid tumors harboring human epidermal growth factor receptor 2 (HER2) activating mutations regardless of tumor histology at 29 investigational sites in 9 countries. First participant was enrolled on 30 Dec 2020, last participant was enrolled on 24 May 2022 and data cut-off (DCO) date was 25 Jan 2023.
Pre-assignment Details: The study consisted of a screening period (up to 28 days), treatment period until progressive disease (PD) and a follow-up period for participants who discontinued study treatment due to PD or other reason. A total of 102 participants received treatment in this study.
Groups:
- Trastuzumab Deruxtecan (T-DXd): Participants harboring tumors with specific HER2 activating mutations received T-DXd 5.4 milligram/kilogram (mg/kg) via intravenous (IV) infusion on Day 1 of each cycle (21 days), every 3 weeks until response evaluation criteria in solid tumors (RECIST) version (v) 1.1 -defined PD, withdrawal of consent, or until any other of the discontinuation criteria was met.
Period: Overall Study
Arm/Group | Trastuzumab Deruxtecan (T-DXd)
Started (Participants assigned to treatment and received treatment) | 102
Completed | 33
Not Completed | 69
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 6
Not completed — Death | 55

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all participants who received at least 1 dose of study treatment.
Groups:
- T-DXd: Participants harboring tumors with specific HER2 activating mutations received T-DXd 5.4 mg/kg via IV infusion on Day 1 of each cycle (21 days), every 3 weeks until RECIST v1.1-defined PD, withdrawal of consent, or until any other of the discontinuation criteria was met.
Arm/Group | T-DXd
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 51
  More than one race | 0
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Overall Response Rate (ORR) as Per RECIST v1.1 Using Independent Central Review (ICR)
Description: Confirmed ORR was defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR), as determined by ICR per RECIST v1.1. A CR was defined as disappearance of all target lesions (TLs) and PR was defined as at least a 30% decrease in the sum of the diameters (dms) of TL, taking as reference the baseline sum of diameters as long as criteria for PD were not met. An ICR of all radiological imaging data was carried out using RECIST v1.1. All images were collected centrally. The imaging scans were reviewed by 2 independent radiologists and were adjudicated, if required.
Time Frame: Tumor scans performed at screening,then every 6 weeks (q6w) +/- 1 week relative to date of first treatment administration until RECIST v1.1 objective PD, withdrawal of consent, or death by any cause, up to DCO date of 25 Jan 2023 (approximately 24 months)
Population: The FAS consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd
Number analyzed (Participants) | 102
percentage of participants | 29.4 [20.8 to 39.3]

2. Secondary Outcome: Duration of Response (DoR) as Per RECIST v1.1 Using ICR and Investigator Assessment
Description: DoR was defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression (date of progression-free survival [PFS] event or censoring - date of first response + 1). The DoR was calculated using Kaplan-Meier technique.
Time Frame: Tumor scans performed at screening, then q6w +/- 1 week relative to the date of first treatment administration until RECIST v1.1 objective PD, withdrawal of consent, or death by any cause, up to DCO date of 25 Jan 2023 (approximately 24 months)
Population: The FAS consisted of all participants who received at least 1 dose of study treatment. Participants with response were evaluated.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | T-DXd
Number analyzed (Participants) | 102
months
  DoR by ICR: number analyzed (Participants) | 30
  DoR by ICR | NA [6.8 to NA] — NA indicates that median and upper limit of confidence interval (CI) were not estimable due to insufficient number of participants with events at study closure.
  DoR by Investigator assessment: number analyzed (Participants) | 33
  DoR by Investigator assessment | 11.0 [6.9 to 18.1]

3. Secondary Outcome: Disease Control Rate (DCR) as Per RECIST v1.1 Using ICR and Investigator Assessment
Description: DCR at 6 weeks was defined as the percentage of participants who had the best objective response (BoR) of confirmed CR or PR, or who had stable disease (SD) (without subsequent cancer therapy), for at least 5 weeks after first dose of study treatment. DCR at 12 weeks was defined as the percentage of patients who had the BoR of confirmed CR or PR, or who had SD (without subsequent cancer therapy), for at least 11 weeks after first dose of study treatment. CR was defined as disappearance of all TL and PR was defined as at least a 30% decrease in sum of the dms of TL, taking as reference the baseline sum of dms as long as criteria for PD were not met. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (>=20% increase in sum of dms of TLs and an absolute increase of >=5 millimeters, taking as reference smallest sum of dms since treatment started including baseline sum of dms). CI was calculated using Clopper-Pearson method.
Time Frame: as for outcome 2
Population: The FAS consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd
Number analyzed (Participants) | 102
percentage of participants
  DCR at 6 weeks by ICR | 75.5 [66.0 to 83.5]
  DCR at 6 weeks by Investigator assessment | 70.6 [60.7 to 79.2]
  DCR at 12 weeks by ICR | 53.9 [43.8 to 63.8]
  DCR at 12 weeks by Investigator assessment | 55.9 [45.7 to 65.7]

4. Secondary Outcome: PFS as Per RECIST v1.1 Using ICR and Investigator Assessment
Description: PFS was defined as the time from first dose of study treatment until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from assigned therapy or received another anti-cancer therapy prior to progression (i.e. date of PFS event or censoring - date of first dose + 1). PFS was calculated using the Kaplan-Meier technique. CI for median PFS derived based on the Brookmeyer-Crowley method.
Time Frame: Tumor scans performed at screening, then q6w +/- 1 week relative to the date of first treatment administration until RECIST v1.1 objective PD or death by any cause, up to DCO date of 25 Jan 2023 (approximately 24 months)
Population: The FAS consisted of all participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd
Number analyzed (Participants) | 102
months
  PFS by ICR | 5.4 [2.7 to 7.1]
  PFS by Investigator assessment | 4.4 [2.8 to 5.6]

5. Secondary Outcome: Percentage of Participants Alive and Progression-Free at 6 and 12 Months as Per RECIST v1.1 Using ICR and Investigator Assessment
Description: Percentage of participants alive and progression-free at 6 and 12 months are reported. It was calculated using the Kaplan-Meier technique. CI for median PFS derived based on the Brookmeyer-Crowley method.
Time Frame: At Months 6 and 12
Population: The FAS consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd
Number analyzed (Participants) | 102
percentage of participants
  PFS rate at 6 months by ICR | 41.4 [30.8 to 51.6]
  PFS rate at 6 months by Investigator assessment | 37.7 [28.1 to 47.2]
  PFS rate at 12 months by ICR | 30.9 [20.6 to 41.8]
  PFS rate at 12 months by Investigator assessment | 26.5 [17.2 to 36.7]

6. Secondary Outcome: Confirmed ORR as Per RECIST v1.1 Using Investigator Assessment
Description: Confirmed ORR was defined as the percentage of participants who had a confirmed CR or PR as determined by investigator per RECIST v1.1. A CR was defined as disappearance of all TLs and PR was defined as >=30% decrease in the sum of the dms of TL, taking as reference the baseline sum of dms as long as criteria for PD were not met.
Time Frame: as for outcome 2
Population: The FAS consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd
Number analyzed (Participants) | 102
percentage of participants | 32.4 [23.4 to 42.3]

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of study treatment administration until death due to any cause regardless of whether the patient withdrew from therapy or received another anti-cancer therapy (i.e. date of death or censoring - date of first dose + 1). OS was calculated using the Kaplan-Meier technique. CI for median OS derived based on the Brookmeyer-Crowley method.
Time Frame: From the date of first treatment administration up to death, approximately 24 months
Population: The FAS consisted of all participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd
Number analyzed (Participants) | 102
months | 10.9 [8.3 to 14.9]

8. Secondary Outcome: Percentage of Participants Alive at 6 and 12 Months
Description: Percentage of participants alive at 6 and 12 months are reported. It was calculated using the Kaplan-Meier technique. CI for median PFS derived based on the Brookmeyer-Crowley method.
Time Frame: At Months 6 and 12
Population: The FAS consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DXd
Number analyzed (Participants) | 102
percentage of participants
  Survival rate at 6 months | 67.6 [57.4 to 75.9]
  Survival rate at 12 months | 46.3 [35.7 to 56.3]

9. Secondary Outcome: Serum Concentrations of T-DXd and Total Anti-HER2 Antibody
Description: Serum samples were collected at specified timepoints to determine serum concentrations of T-DXd and total anti-HER2 antibody.
Time Frame: Pre-infusion and 15 minutes post-infusion in Cycles 1, 2 and 4 and 5 hours post-infusion in Cycle 1 (each cycle 21 days)
Population: The Pharmacokinetic (PK) Analysis set consisted of all participants who received at least 1 dose of study treatment and had at least 1 post-dose evaluable PK data point. The population was defined by the study pharmacokineticist and the statistician prior to any PK analyses being performed. Only those participants with data available are reported.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mL)
Arm/Group | T-DXd
Number analyzed (Participants) | 100
microgram/milliliter (mL)
  T-DXd: Cycle 1: Pre-infusion: number analyzed (Participants) | 1
  T-DXd: Cycle 1: Pre-infusion | NA (NA) — Mean was <lower limit of quantification (LLOQ). LLOQ was 400 nanogram (ng)/mL.
  T-DXd: Cycle 1: 15 minutes post-infusion: number analyzed (Participants) | 96
  T-DXd: Cycle 1: 15 minutes post-infusion | 116.5 (50.8)
  T-DXd: Cycle 1: 5 hours post-infusion: number analyzed (Participants) | 98
  T-DXd: Cycle 1: 5 hours post-infusion | 115.4 (30.5)
  T-DXd: Cycle 2: Pre-infusion: number analyzed (Participants) | 91
  T-DXd: Cycle 2: Pre-infusion | 11.2 (74.1)
  T-DXd: Cycle 2: 15 minutes post-infusion: number analyzed (Participants) | 93
  T-DXd: Cycle 2: 15 minutes post-infusion | 132.2 (101.5)
  T-DXd: Cycle 4: Pre-infusion: number analyzed (Participants) | 59
  T-DXd: Cycle 4: Pre-infusion | 7.7 (9.1)
  T-DXd: Cycle 4: 15 minutes post-infusion: number analyzed (Participants) | 59
  T-DXd: Cycle 4: 15 minutes post-infusion | 121.7 (40.1)
  Total anti-HER2 antibody: Cycle 1: Pre-infusion: number analyzed (Participants) | 9
  Total anti-HER2 antibody: Cycle 1: Pre-infusion | NA (NA) — Mean was <LLOQ. LLOQ was 400 ng/mL.
  Total anti-HER2 antibody: Cycle 1: 15 minutes post-infusion: number analyzed (Participants) | 97
  Total anti-HER2 antibody: Cycle 1: 15 minutes post-infusion | 123.8 (52.8)
  Total anti-HER2 antibody: Cycle 1: 5 hours post-infusion: number analyzed (Participants) | 97
  Total anti-HER2 antibody: Cycle 1: 5 hours post-infusion | 122.1 (42.1)
  Total anti-HER2 antibody: Cycle 2: Pre-infusion: number analyzed (Participants) | 88
  Total anti-HER2 antibody: Cycle 2: Pre-infusion | 6.2 (12.4)
  Total anti-HER2 antibody: Cycle 2: 15 minutes post-infusion: number analyzed (Participants) | 94
  Total anti-HER2 antibody: Cycle 2: 15 minutes post-infusion | 144.4 (115.4)
  Total anti-HER2 antibody: Cycle 4: Pre-infusion: number analyzed (Participants) | 58
  Total anti-HER2 antibody: Cycle 4: Pre-infusion | 9.9 (5.7)
  Total anti-HER2 antibody: Cycle 4: 15 minutes post-infusion: number analyzed (Participants) | 59
  Total anti-HER2 antibody: Cycle 4: 15 minutes post-infusion | 122.1 (37.3)

10. Secondary Outcome: Serum Concentrations of Deruxtecan (MAAA-1181a)
Description: Serum samples were collected at specified timepoints to determine serum concentrations of MAAA-1181a.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | T-DXd
Number analyzed (Participants) | 100
ng/mL
  MAAA-1181a: Cycle 1: Pre-infusion: number analyzed (Participants) | 0
  MAAA-1181a: Cycle 1: 15 minutes post-infusion: number analyzed (Participants) | 99
  MAAA-1181a: Cycle 1: 15 minutes post-infusion | 4.7 (2.9)
  MAAA-1181a: Cycle 1: 5 hours post-infusion: number analyzed (Participants) | 95
  MAAA-1181a: Cycle 1: 5 hours post-infusion | 10.5 (5.1)
  MAAA-1181a: Cycle 2: Pre-infusion: number analyzed (Participants) | 90
  MAAA-1181a: Cycle 2: Pre-infusion | 0.2 (0.1)
  MAAA-1181a: Cycle 2: 15 minutes post-infusion: number analyzed (Participants) | 94
  MAAA-1181a: Cycle 2: 15 minutes post-infusion | 2.2 (1.5)
  MAAA-1181a: Cycle 4: Pre-infusion: number analyzed (Participants) | 57
  MAAA-1181a: Cycle 4: Pre-infusion | 0.3 (0.2)
  MAAA-1181a: Cycle 4: 15 minutes post-infusion: number analyzed (Participants) | 58
  MAAA-1181a: Cycle 4: 15 minutes post-infusion | 1.5 (0.9)

11. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) to T-DXd
Description: Blood samples were collected to evaluate the presence of ADAs for T-DXd using validated assays. ADA prevalence was defined as the percentage of participants with positive ADA result at any time, baseline or post-baseline. ADA incidence was defined as the percentage of participants who were evaluable for ADA and were treatment-emergent ADA-positive. Treatment-emergent ADA was defined as either treatment-induced (baseline ADA negative, post-baseline ADA positive) or treatment-boosted ADA. Treatment-boosted ADA was defined as baseline positive ADA titer that was boosted to >=2 fold during the study period. Persistently positive was defined as >=2 post-baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. Transiently positive was defined as having >=1 post baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: Up to approximately 24 months
Population: Participants in the ADA-evaluable set consisted of all participants in the Safety Analysis set (SAF- All participants who received at least 1 dose of study treatment) with a non-missing baseline ADA result and at least 1 non-missing post-baseline ADA result.
Measure: Number; unit: percentage of participants
Arm/Group | T-DXd
Number analyzed (Participants) | 96
percentage of participants
  ADA positive at any visit (ADA prevalence) | 2.1
  ADA incidence | 0
  Treatment-emergent ADA positive | 0
  Treatment-boosted ADA positive | 0
  Persistently positive ADA | 0
  Transiently positive ADA | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from start of first dose of study treatment up to and including 47 days following the date of last dose of study treatment or before the initiation of first subsequent anti-cancer therapy following discontinuation of study treatment (whichever occurred first), up to DCO date of 25 Jan 2023 (approximately 24 months)
Description: The SAF consisted of all participants who received at least 1 dose of study treatment.
Groups:
- T-DXd: Description (Arm-group)
Arm/Group | T-DXd
All-Cause Mortality (participants affected / at risk) | 58/102
Serious Adverse Events (participants affected / at risk) | 36/102
Other Adverse Events (participants affected / at risk) | 96/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DXd (N=102)
Sepsis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 2 (2)
Complication associated with device (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2)
Biliary tract infection (Infections and infestations) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DXd (N=102)
Alanine aminotransferase increased (Investigations) | 14 (18)
Aspartate aminotransferase increased (Investigations) | 18 (21)
Neutrophil count decreased (Investigations) | 15 (26)
Platelet count decreased (Investigations) | 13 (18)
Decreased appetite (Metabolism and nutrition disorders) | 24 (24)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Headache (Nervous system disorders) | 8 (8)
Anaemia (Blood and lymphatic system disorders) | 35 (41)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Abdominal pain (Gastrointestinal disorders) | 12 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
Ascites (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 18 (24)
Diarrhoea (Gastrointestinal disorders) | 28 (31)
Dyspepsia (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 49 (66)
Stomatitis (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 13 (15)
Asthenia (General disorders) | 19 (20)
Fatigue (General disorders) | 31 (39)
Malaise (General disorders) | 7 (7)
Oedema peripheral (General disorders) | 9 (9)
Neutropenia (Blood and lymphatic system disorders) | 6 (7)
Pyrexia (General disorders) | 11 (15)
COVID-19 (Infections and infestations) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT04639219/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT04639219/SAP_001.pdf